CLINICAL TRIAL: NCT04725422
Title: CHronic Nonbacterial Osteomyelitis International Registry (CHOIR)
Brief Title: CHronic Nonbacterial Osteomyelitis International Registry
Acronym: CHOIR
Status: Recruiting | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Boston Children's Hospital, Boston, MA, USA (Other); Hospital for Special Surgery, New York (Other); Joseph M Sanzari Children's Hospital, Hackensack University Medical Center, Hackensack, NJ, USA (Unknown); Riley Children's Hospital, Indianapolis, IN, USA (Unknown); University of North Carolina, Chapel Hill, NC, USA (Unknown); Royal Children's Hospital (Other); Hacettepe University (Other); Bambino Gesù Children's Hospital, Rome, Italy (Unknown); University of British Columbia, Vancouver, BC, Canada (Unknown); Meyer Children's Hospital, Florence, Italy (Unknown); Mansoura University (Other); University of Utah, Salt Lake City, UT, USA (Unknown); University of Iowa Carver College of Medicine, Iowa City, IA, USA (Unknown); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Palacky University Olomouc Institute of Molecular and Translational Medicine, Olomouc, Czechia (Unknown); Alder Hey Children's NHS Foundation Trust (Other); University of Calgary, Calgary, Alberta, Canada (Unknown)
Responsible Party: Principal Investigator, Yongdong (Dan) Zhao, Principle Investigator, Seattle Children's Hospital
Other Study IDs: 1232
Record Dates: First submitted 2021-01-18; First posted 2021-01-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Chronic Nonbacterial Osteomyelitis; Chronic Recurrent Multifocal Osteomyelitis
MeSH Terms: conditions — Chronic recurrent multifocal osteomyelitis | interventions — Methotrexate; Sulfasalazine; Leflunomide; Pamidronate; Zoledronic Acid; Etanercept; Adalimumab; Certolizumab Pegol; Infliximab; golimumab; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- disease modifying anti-rheumatic drug, DMARD: 1. Methotrexate 1 mg/kg (max 25 mg) PO or SQ weekly
  2. Sulfasalazine 30 mg/kg (max 1000 mg) PO twice daily
  3. Leflunomide 10-20 mg PO daily
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Leflunomide
- tumor necrosis factor inhibitor, TNFi: 1. Adalimumab (subcutaneous) 10-40 mg SQ every other week
  2. Etanercept (subcutaneous) 12.5-50 mg SQ every week
  3. Infliximab (intravenous) 10 mg/kg (max 1000 mg) i.v. at week 0,2, 6 then every 4 weeks
  4. Golimumab (subcutaneous or intravenous) 2 mg/kg (max 200 mg) at every 4 weeks
  Interventions: Drug: Etanercept; Drug: Adalimumab; Drug: Certolizumab; Drug: Infliximab; Drug: Golimumab
- bisphosphonate: 1. Pamidronate 1 mg/kg (max 90 mg) (intravenous)*:
     Option 1: every month Option 2: 3 consecutive days every 3 months
  2. Zoledronic acid 0.0125-0.05 mg/kg (max 4mg) (intravenous): every 3-6 months. * Both options may use lower dose of 0.5 mg/kg at the initiation of the treatment. All options allow concurrent use of NSAIDs.
  Interventions: Drug: Pamidronate; Drug: Zoledronic acid
- non-steroidal anti-inflammatory drugs: 1. Naproxen 10 mg/kg (max 500 mg) PO twice daily
  2. Indomethacin 1 mg/kg (max daily dose 150 mg) PO twice or three times daily
  3. Meloxicam 0.1-0.3 mg/kg (max 15 mg) PO daily
  4. Piroxicam 10-20 mg PO daily
  5. Ibuprofen 10 mg/kg (max 800 mg) PO 3-4 times daily
  Interventions: Drug: NSAID

INTERVENTIONS:
Drug: Methotrexate — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Groups: disease modifying anti-rheumatic drug, DMARD
Drug: Sulfasalazine — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Other Names: Azulfidine
  Groups: disease modifying anti-rheumatic drug, DMARD
Drug: Leflunomide — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Other Names: areva
  Groups: disease modifying anti-rheumatic drug, DMARD
Drug: Pamidronate — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Other Names: Aredia
  Groups: bisphosphonate
Drug: Zoledronic acid — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Groups: bisphosphonate
Drug: Etanercept — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Other Names: enbrel
  Groups: tumor necrosis factor inhibitor, TNFi
Drug: Adalimumab — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Other Names: humira
  Groups: tumor necrosis factor inhibitor, TNFi
Drug: Certolizumab — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Other Names: cimzia
  Groups: tumor necrosis factor inhibitor, TNFi
Drug: Infliximab — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Other Names: remicade, inflectra
  Groups: tumor necrosis factor inhibitor, TNFi
Drug: Golimumab — second-line treatment for children with CNO/CRMO after failure to respond to NSAIDs
  Other Names: simponi
  Groups: tumor necrosis factor inhibitor, TNFi
Drug: NSAID — first-line treatment
  Groups: non-steroidal anti-inflammatory drugs

SUMMARY:
The objective of the study is to establish a prospective disease registry for chronic recurrent multifocal osteomyelitis (CRMO)/chronic nonbacterial osteomyelitis (CNO) in order to investigate the natural history of the disease and the responses of patients to different clinical managements over 10 years.

DETAILED DESCRIPTION:
Chronic nonbacterial osteomyelitis (CNO) is an autoinflammatory bone disease that mainly affects children and adolescents. Clinical presentations range from mild and sometimes limited unifocal disease to severe, chronically active or recurrent inflammation of multiple bones. The latter is referred to as chronic recurrent multifocal osteomyelitis (CRMO). Here we will use the term "CNO" to refer to the entire spectrum of this disease. CNO can be complicated by vertebral compression fractures, kyphosis, and leg length discrepancy when it is not recognized early or treated adequately. The diagnosis of CNO is made by excluding alternatives in the differential diagnosis including malignancy (leukemia, lymphoma, and primary or metastatic bone tumors), Langerhans cell histiocytosis, and infection. Clinical assessment in conjunction with serum inflammatory parameters and imaging studies, particularly magnetic resonance imaging (MRI), are crucial for the diagnosis and monitoring of disease activity of CNO1.

Because of significant variation in clinical treatment practices among pediatric rheumatologists, standardized treatment regimens (consensus treatment plans, CTPs) have been developed within the Childhood Arthritis and Rheumatology Research Alliance (CARRA), a North American organization comprised of pediatric rheumatologists and researchers, for CNO patients with an NSAID-refractory course and/or with active spinal lesions2. These CTPs provide an opportunity for pediatric rheumatologists to conduct comparative effectiveness research on CNO through prospective data collection. CRMO/CNO workgroup is comprised of pediatric rheumatologists from North America as well as international colleagues who are interested in collaborating in CNO research. Furthermore, risk factors of severe disease have been described by Wipff et al. based on a large retrospective cohort study3. Their results may be validated by an independent prospective cohort study. To date, there has been only one prospective study on CNO since its first description in 19724. Therefore, we propose to establish this international registry of patients with CNO to accomplish above goals. Long-term outcomes of CNO remains unknown due to the lack of prospective study. It has been estimated that at least 50% of CNO patients continue to need medications for CNO during adulthood. Our study will collect the clinical data and provide valuable data to characterize the long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* - Age at enrollment is equal to or younger than 21 years of age
* Presence of bone edema on STIR or T2 fat saturation sequence on MRI within 12 weeks of enrollment
* Whole body imaging evaluation (either WB MRI or bone scintigraphy)
* Bone biopsy to exclude infection or malignancy unless bone lesions follow typical distribution or there is IBD, psoriasis, or palmar plantar pustulosis

Exclusion Criteria:

* - History of or current malignancy
* Current infectious osteomyelitis
* Contraindication to the selected treatment agent

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with a diagnosis of CNO/CRMO who have failed NSAIDs and/or with active spinal lesion
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2050-08 (Estimated)

PRIMARY OUTCOMES:
The change of CNO disease activity score | 3-6 months
  Disease activity score is calculated as the sum of number of clinical lesion count, patient global assessment (0-10), physician global assessment (0-10)

SECONDARY OUTCOMES:
Total number of CNO lesions on MRI | 3-6 months
  The total number of CNO lesions from MRI as previously described (Zhao, et al. J Rheum 2019) will be used to monitor response in a subset
Safety monitoring | 5 years
  Serious adverse events including infections that require IV antibiotics, malignancy, hematological, hepatic, dermatological side effects will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao Y, Wu EY, Oliver MS, Cooper AM, Basiaga ML, Vora SS, Lee TC, Fox E, Amarilyo G, Stern SM, Dvergsten JA, Haines KA, Rouster-Stevens KA, Onel KB, Cherian J, Hausmann JS, Miettunen P, Cellucci T, Nuruzzaman F, Taneja A, Barron KS, Hollander MC, Lapidus SK, Li SC, Ozen S, Girschick H, Laxer RM, Dedeoglu F, Hedrich CM, Ferguson PJ; Chronic Nonbacterial Osteomyelitis/Chronic Recurrent Multifocal Osteomyelitis Study Group and the Childhood Arthritis and Rheumatology Research Alliance Scleroderma, Vasculitis, Autoinflammatory and Rare Diseases Subcommittee. Consensus Treatment Plans for Chronic Nonbacterial Osteomyelitis Refractory to Nonsteroidal Antiinflammatory Drugs and/or With Active Spinal Lesions. Arthritis Care Res (Hoboken). 2018 Aug;70(8):1228-1237. doi: 10.1002/acr.23462. Epub 2018 Jul 12. PMID 29112802
- [Background] Zhao Y, Ferguson PJ. Chronic Nonbacterial Osteomyelitis and Chronic Recurrent Multifocal Osteomyelitis in Children. Pediatr Clin North Am. 2018 Aug;65(4):783-800. doi: 10.1016/j.pcl.2018.04.003. PMID 30031498
- [Background] Oliver M, Lee TC, Halpern-Felsher B, Murray E, Schwartz R, Zhao Y; CARRA SVARD CRMO/CNO workgroup. Disease burden and social impact of pediatric chronic nonbacterial osteomyelitis from the patient and family perspective. Pediatr Rheumatol Online J. 2018 Dec 14;16(1):78. doi: 10.1186/s12969-018-0294-1. PMID 30547806
- [Background] Beck C, Morbach H, Beer M, Stenzel M, Tappe D, Gattenlohner S, Hofmann U, Raab P, Girschick HJ. Chronic nonbacterial osteomyelitis in childhood: prospective follow-up during the first year of anti-inflammatory treatment. Arthritis Res Ther. 2010;12(2):R74. doi: 10.1186/ar2992. PMID 20433730
- [Background] Girschick H, Finetti M, Orlando F, Schalm S, Insalaco A, Ganser G, Nielsen S, Herlin T, Kone-Paut I, Martino S, Cattalini M, Anton J, Mohammed Al-Mayouf S, Hofer M, Quartier P, Boros C, Kuemmerle-Deschner J, Pires Marafon D, Alessio M, Schwarz T, Ruperto N, Martini A, Jansson A, Gattorno M; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Eurofever registry. The multifaceted presentation of chronic recurrent multifocal osteomyelitis: a series of 486 cases from the Eurofever international registry. Rheumatology (Oxford). 2018 Jul 1;57(7):1203-1211. doi: 10.1093/rheumatology/key058. PMID 29596638
- [Background] Voit AM, Arnoldi AP, Douis H, Bleisteiner F, Jansson MK, Reiser MF, Weckbach S, Jansson AF. Whole-body Magnetic Resonance Imaging in Chronic Recurrent Multifocal Osteomyelitis: Clinical Longterm Assessment May Underestimate Activity. J Rheumatol. 2015 Aug;42(8):1455-62. doi: 10.3899/jrheum.141026. Epub 2015 May 15. PMID 25979713
- [Background] Wu EY, Oliver M, Scheck J, Lapidus S, Akca UK, Yasin S, Stern SM, Insalaco A, Pardeo M, Simonini G, Marrani E, Wang X, Huang B, Kovalick LK, Rosenwasser N, Casselman G, Liau A, Shao Y, Yang C, Mosa DM, Tucker L, Girschick H, Laxer RM, Akikusa JD, Hedrich CM, Onel K, Dedeoglu F, Twilt M, Ferguson PJ, Ozen S, Zhao Y. Feasibility of Conducting Comparative Effectiveness Research and Validation of a Clinical Disease Activity Score for Chronic Nonbacterial Osteomyelitis. J Rheumatol. 2023 Oct;50(10):1333-1340. doi: 10.3899/jrheum.2022-1323. Epub 2023 Jul 1. PMID 37399459

DOCUMENTS (2):
  • Study Protocol (2023-11-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT04725422/Prot_000.pdf
  • Informed Consent Form (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT04725422/ICF_001.pdf